CLINICAL TRIAL: NCT06871774
Title: Comparative Efficacy of Single vs. Dual Perclose Devices for Large-Bore Access Closure in Transcatheter Aortic Valve Replacement: A Randomized Controlled Trial
Brief Title: Comparison of Single vs. Dual Perclose Devices for Large-Bore Access Closure in TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00124842
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: aortic valve diseases; Perclose device; arteriotomy
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Single Device (Experimental): A single Perclose device will be used for pre-closure of the vascular access site, with manual pressure and up to two additional devices used as needed to achieve hemostasis.
  Interventions: Device: Single Perclose Pro vascular closure device
- Two device (Active Comparator): Two Perclose devices will be used for pre-closure of the vascular access site, with manual pressure and an additional device used as needed to achieve hemostasis.
  Interventions: Device: Dual Perclose vascular closure device

INTERVENTIONS:
Device: Single Perclose Pro vascular closure device — Use of a single Perclose device for pre-closure of vascular access site after removal of TAVR sheath.
  Arms: Single Device
Device: Dual Perclose vascular closure device — Use of two Perclose devices for pre-closure of vascular access site after removal of TAVR sheath.
  Arms: Two device

SUMMARY:
This study will compare the use of one Perclose device to the usual approach of two devices for pre-closure during Transcatheter Aortic Valve Replacement (TAVR). The study will compare the time it takes for bleeding to stop using the different closure approaches. The study will also compare complications when using one Perclose device versus two.

DETAILED DESCRIPTION:
This single-center randomized trial compares single versus dual Perclose devices for pre-closure of vascular access for Transcatheter Aortic Valve Replacement (TAVR) and investigation will evaluate the efficacy and performance of these two pre-closure approaches. The study will provide valuable insights into optimizing pre-closure techniques, potentially enhancing patient outcomes and reducing complications associated with Transcatheter Aortic Valve Replacement (TAVR) procedures. The trial will aim to enroll patients undergoing TAVR, with an an equal number of patients randomized to each pre-closure strategy arm.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 or older
* Transfemoral transcatheter aortic valve replacement (TAVR)
* Implantation of CoreValve replacement valve
* Access using 14 French sheaths
* English speaking

Exclusion Criteria:

* Alternative Access Routes: Patients undergoing transcatheter aortic valve replacement (TAVR) via alternative access routes such as subclavian access or transapical access.
* Planned Surgical Cut-Down: Patients planned for surgical cut-down procedures rather than percutaneous access.
* Vascular Access Complications: Patients with known vascular complications at the femoral access site, such as residual hematoma, recent femoral arteriotomy or venotomy within the past 10 days, history of significant vascular complications or prior intravascular closure device use within the previous 30 days.
* Arterial or Venous Issues: Patients with small femoral arteries or veins (<5 mm in diameter), patients with access sites located in vascular grafts.
* Body Composition: Patients with BMI >35
* Cardiac Vasculature: Patients with excess calcification of vessels as determined by echocardiography and/or CT angiography
* Infection or Inflammation: Active systemic or cutaneous infection or inflammation in the vicinity of the groin.
* Coagulation and Hematological Disorders: Known history of bleeding diathesis, coagulopathy, hypercoagulability, or platelet count <100,000 cells/mm³. Pre-existing immunodeficiency disorder or chronic use of high-dose systemic steroids.
* Severe Morbidity: Severe co-existing morbidities with a life expectancy less than 12 months.
* Mobility Issues: Patients unable to routinely walk at least 20 feet without assistance.
* Recent Anticoagulation: Use of low molecular weight heparin (LMWH) within 8 hours before or after the procedure.
* Pregnancy and Lactation: Pregnant or lactating women.
* Incompatible Procedure Plan: Patients receiving the Edwards Sapien valve (Edwards Lifesciences, Irvine, CA)
* Contraindications: Patients with contraindications for the use of Perclose device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Vascular Complications | Day 5 post-procedure
  Number of subjects in each group experiencing major or minor vascular complications directly related to the TAVR procedure occurring during the index hospitalization.
Number of Patients With Life-threatening bleeding | Hour 24 post-procedure
  Number of subjects in each group experiencing any bleeding event related to the TAVR procedure that is life-threatening within 24 hours post-procedure.
Number of Patients With Major or Minor Bleeding Complications Without Life-Threatening Condition | Hour 24 post-procedure
  Number of subjects in each group experiencing bleeding complications related to the TAVR procedure that do not meet the criteria for life-threatening bleeding but still result in significant clinical concern within 24 hours of the index procedure.
Time to Hemostasis | 1 hour post procedure
  For each subject, time elapsed from initial deployment of the initial one or two Perclose devices (depending on assigned group) to complete hemostasis of the femoral access site. Measured in seconds.

SECONDARY OUTCOMES:
Additional Closure Device Use | Hour 24 post-procedure
  Number of subjects requiring use of additional closure devices beyond the initial closure strategy required to achieve hemostasis at the femoral access site within 24 hours post-procedure. The number and type of devices will be recorded for each subject.
In-Hospital Serious Vascular Complications Requiring Percutaneous or Surgical Interventions | Day 5 post-procedure
  Number of subjects in each group experiencing severe vascular complications that necessitate either percutaneous procedures or surgical interventions during the index hospitalization.
Number of Patients With Limb Ischemia Related to TAVR During Index Admission | Day 5 post-procedure
  Number of subjects in each group experiencing significant peripheral ischemia related to the arteriotomy closure between the TAVR procedure and discharge.
Limb Ischemia Related to TAVR | Day 30 post-procedure
  Number of subjects in each group experiencing significant peripheral ischemia related to the arteriotomy closure monitored within 30 days post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Q Allaqaband, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No